CLINICAL TRIAL: NCT01814670
Title: Treatment With Botulinum Toxin Type A (BOTOX®) in Chinese Patients With Moderate to Severe Frown Lines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP-BTXC-12-001
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Results first posted 2015-09-01 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Glabellar Rhytides
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- botulinum toxin Type A (Experimental): 20 units botulinum toxin Type A (total dose) injected into frown lines on Day 1.
  Interventions: Biological: botulinum toxin Type A

INTERVENTIONS:
Biological: botulinum toxin Type A — 20 units botulinum toxin Type A (total dose) injected into frown lines on Day 1.
  Other Names: BOTOX®; onabotulinumtoxinA

SUMMARY:
A study to evaluate safety and efficacy of treatment with botulinum toxin Type A (BOTOX®) in Chinese patients with moderate to severe frown lines (Glabellar Rhytides) previously treated with facial laser resurfacing.

ELIGIBILITY:
Inclusion Criteria:

* moderate or severe frown lines
* facial laser treatment between 4 to 8 weeks prior to Day 1

Exclusion Criteria:

* previous use of botulinum toxin for any indication
* diagnosis of myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis
* microdermabrasion or superficial peels, permanent make-up to the brow and forehead area within the last 3 months
* facial cosmetic procedures within the last 6 Months
* treatment to forehead, brow, nose or midface areas with any filler within the last 12 months
* use of a new topical skin care product within 1 month of the screening
* any prior forehead or periorbital surgery or brow lift
* deep dermal scarring, excessively thick sebaceous skin, and/ or loss of skin elasticity
* any facial skin infection or unhealed skin lesion
* pregnant or breast-feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 185 (Actual)
Dates: Start 2013-03-06 (Actual); Primary Completion 2014-07-31 (Actual); Study Completion 2014-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Beijing, China

REFERENCES:
- [Background] Wu Y, Lu Z, Xie Y, Zhang W, Chen X, Shi Y, Li Q, Halstead M, Rogers JD, Silberberg M. OnabotulinumtoxinA treatment of moderate to severe glabellar lines in Chinese subjects after laser therapy: A prospective, open-label, noncomparative study. J Cosmet Laser Ther. 2018 Oct;20(5):278-286. doi: 10.1080/14764172.2017.1406604. Epub 2018 Mar 2. PMID 29498553

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin Type A
Started | 185
Completed | 173
Not Completed | 12
Not completed — Protocol Violation | 12

BASELINE CHARACTERISTICS:
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 185
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.8 (8.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With a ≥ 1-Grade Improvement From Day 1 in the Investigator Assessed Facial Wrinkle Scale of Glabellar Rhytides at Maximum Contraction
Description: The Investigator assessed the severity of the subject's glabellar rhytides at maximum contraction using the 4-point Facial Wrinkle Scale: 0=none, 1=mild, 2=moderate or 3=severe. The percentage of subjects with a ≥ 1-grade improvement from Day 1 is reported.
Time Frame: Day 1, Day 30
Population: Intent-to-Treat: all eligible subjects enrolled in the study who received study treatment (BOTOX®) at Day 1
Measure: Number; unit: Percentage of Subjects
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 173
Percentage of Subjects | 97.1

2. Secondary Outcome: Percentage of Subjects With a ≥ 1-Grade Improvement From Day 1 in the Investigator Assessed Facial Wrinkle Scale of Glabellar Rhytides at Maximum Contraction
Description: as for outcome 1
Time Frame: Day 1, Day 14, Day 90, Day 120
Population: Intent-to-Treat: all eligible subjects enrolled in the study who received study treatment (BOTOX®) at Day 1
Measure: Number; unit: Percentage of Subjects
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 173
Percentage of Subjects
  Day 14 | 97.1
  Day 90 | 90.2
  Day 120 | 81.5

3. Secondary Outcome: Percentage of Subjects With a ≥ 1-Grade Improvement From Day 1 in the Subject Assessed Facial Wrinkle Scale of Glabellar Rhytides at Maximum Contraction
Description: The subject assessed the severity of his/her glabellar rhytides at maximum contraction using the 4-point Facial Wrinkle Scale: 0=none, 1=mild, 2=moderate or 3=severe. The percentage of subjects with a ≥ 1-grade improvement from Day 1 is reported.
Time Frame: Day 1, Day 14, Day 30, Day 90, Day 120
Population: Intent-to-Treat: all eligible subjects enrolled in the study who received study treatment (BOTOX®) at Day 1 and had data at the noted time point
Measure: Number; unit: Percentage of Subjects
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 173
Percentage of Subjects
  Day 14 | 90.1
  Day 30 | 93.1
  Day 90 | 81.5
  Day 120 | 72.3

4. Secondary Outcome: Percentage of Subjects With a ≥ 1-Grade Improvement From Day 1 in the Investigator Assessed Facial Wrinkle Scale of Glabellar Rhytides at Rest
Description: The Investigator assessed the severity of the subject's glabellar rhytides at rest using the 4-point Facial Wrinkle Scale: 0=none, 1=mild, 2=moderate or 3=severe. The percentage of subjects with a ≥ 1-grade improvement from Day 1 is reported.
Time Frame: Day 1, Day 14, Day 30, Day 90, Day 120
Population: Intent-to-Treat: all eligible subjects enrolled in the study who received study treatment (BOTOX®) at Day 1
Measure: Number; unit: Percentage of Subjects
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 173
Percentage of Subjects
  Day 14 | 62.7
  Day 30 | 65.7
  Day 90 | 65.7
  Day 120 | 62.7

5. Secondary Outcome: Percentage of Subjects With a ≥ 1-Grade Improvement From Day 1 in the Subject Assessed Facial Wrinkle Scale of Glabellar Rhytides at Rest
Description: The Subject assessed the severity of his/her glabellar rhytides at rest using the 4-point Facial Wrinkle Scale: 0=none, 1=mild, 2=moderate or 3=severe. The percentage of subjects with a ≥ 1-grade improvement from Day 1 is reported.
Time Frame: Day 1, Day 14, Day 30, Day 90, Day 120
Population: Intent-to-Treat: all eligible subjects enrolled in the study who received study treatment (BOTOX®) at Day 1
Measure: Number; unit: Percentage of Subjects
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 173
Percentage of Subjects
  Day 14 | 59.9
  Day 30 | 58.4
  Day 90 | 50.9
  Day 120 | 49.1

ADVERSE EVENTS:
Description: The Safety Population was used to assess adverse events (AEs) and serious adverse events (SAEs).
Arm/Group | Botulinum Toxin Type A
Serious Adverse Events (participants affected / at risk) | 0/185
Other Adverse Events (participants affected / at risk) | 0/185

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.